CLINICAL TRIAL: NCT04290247
Title: Non-inferiority of Ultrasound for the Diagnosis of Upper Extremity Fractures in Children
Acronym: FRUSKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Principal Investigator, David Troxler, Principal Investigator, University Children's Hospital Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UKBB-2020/001; 2020-00032 (Registry Identifier: BASEC)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Fracture Diagnosis by Ultrasound Compared to X-ray
Keywords: Pediatric; Ultrasound; X-ray; Fracture; Diagnosis
MeSH Terms: conditions — Fractures, Bone; Disease | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Ultrasound before X-ray for all included patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound + X-ray (Experimental): Ultrasound first then x-ray examination
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound imaging for fracture diagnosis before conventional X-ray

SUMMARY:
This study evaluates the sensitivity of Ultrasound for Diagnostic of Fractures of the upper extremity compared to conventional x-ray in Children 0-18.

DETAILED DESCRIPTION:
Fractures of the upper extremity are common in children. Approximately 200 children with a suspected upper extremity fracture are treated every month in the paediatric emergency room (pER) of the University Hospital of Basel-Stadt and Basel-Land (UKBB).

If a fracture is suspected in the emergency room, two separate X-ray images have to be obtained to diagnose or exclude a fracture, according to the current standard operating procedure (SOP). This procedure has several disadvantages as X-ray imaging exposes children to radiation and transfer to the X-ray facility is time-consuming. Depending on the suspected fracture, the broken limb needs to be positioned for the two separate perspectives of the images, resulting in pain.

Furthermore, this procedure is time-consuming as the work routine of the attending emergency room physician is interrupted once the child is sent to the imaging facility and then returns to the emergency room after the procedure. The time between the request of the examination and interpretation of the results is called therapeutic turnaround time or brain-to-brain time.

X-ray images are interpreted by the pER paediatrician, and treatment is based upon this interpretation. A secondary reading by a paediatric radiologist for quality control is only done later on. This procedure has been adopted by several hospitals internationally.

X-ray interpretation by pER paediatricians has been evaluated by various studies, and the accuracy compared to paediatric radiologist interpretation is around 90% in most studies, with extremes ranging from 84% to 99%. In the past few years, ultrasound diagnosis of upper extremity fractures in adults and children has been studied. However, the evidence of its effectiveness is still limited, and its application in routine care is uncommon.

Ultrasound has several advantages over X-ray imaging. It does not expose patients to radiation; devices are mobile, the examination can be performed in the child's preferred antalgic position without moving the affected limb, it is always available, and it can be executed directly by an emergency room physician.

We aim to demonstrate that ultrasound is at least as sensitive as X-ray imaging and is thus non-inferior to the standard-of-care diagnostics with X-ray.

Secondary outcomes include pain and time necessary for ultrasound vs X-ray If non-inferiority can be confirmed in this study, we expect a change in SOPs to replace initial X ray imaging by sonographic fracture diagnosis for simple fractures of the upper-extremity long bones.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency room of the UKBB with a history of acute trauma to the upper extremities and suspected fracture of a long bone
* Age 0-18 years

Exclusion Criteria:

* Patient needing immediate medical attention (triage score 1 or 2)
* Severely displaced or open fractures
* Patient with neurovascular compromise distally to the suspected fracture.
* Patient with imaging studies obtained prior to the emergency room visit
* Patient with prior fracture of the affected area
* Patient with known allergy to ultrasound gel.
* Patient with suspected 'battered child' diagnosis.
* Unavailability of a study investigator able to perform the ultrasound examination within a reasonable time frame (15 min; see also 3.2).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 428 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 1 year
  Sensitivity of Ultrasound diagnostic compared to X-ray

SECONDARY OUTCOMES:
Pain level | 1 year
  Pain during Ultrasound imaging compared to X-ray imaging
Time | 1 year
  Time necessary for Ultrasound imaging compared to X-ray imaging
Displacement | 2 years
  Specification of Displacement measures by Ultrasound imaging compared to X-ray imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- University Childrens Hospital for both Basel cantons, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Troxler D, Sanchez C, de Trey T, Mayr J, Walther M. Non-Inferiority of Point-of-Care Ultrasound Compared to Radiography to Diagnose Upper Extremity Fractures in Children. Children (Basel). 2022 Sep 30;9(10):1496. doi: 10.3390/children9101496. PMID 36291432